CLINICAL TRIAL: NCT05266170
Title: The Effect of EX1 Training on Muscle Activity, Heart Rate, and Respiratory Metabolic Energy Consumption Rate in Normal Adults
Brief Title: The Effect of EX1 Training in Normal Adults
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-12-153
Record Dates: First submitted 2022-02-06; First posted 2022-03-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-01

CONDITIONS: Aerobic Exercises; Anaerobic Exercises

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal adults: aerobic and anaerobic exercises
  Interventions: Device: aerobic and anaerobic exercises

INTERVENTIONS:
Device: aerobic and anaerobic exercises — [aerobic]
  1. Aerobic treadmill walking program without EX1
  2. Aerobic treadmill walking program with EX1
  3. High-intensity interval exercise (HIIT) program with EX1
  [anaerobic]
  1. Fitness exercise program with EX1

SUMMARY:
In this study, when performing aerobic and anaerobic exercise with EX1 applied to normal adults between the ages of 19 and 65. The purpose of this study was to determine the effect on the muscle activity of the trunk and lower extremities compared with and without EX1.

DETAILED DESCRIPTION:
In this study, aerobic exercise and anaerobic exercise for normal adults were divided into two visits for a total. For aerobic exercise, the investigators compared the aerobic treadmill walking program without EX1 [30 minutes of moderate (64-76% HRmax, 12-14 of RPE) aerobic treadmill walking, 40 minutes including warm-up and cool-down times], the aerobic treadmill walking program with EX1 [30 minutes of moderate (64-76% HRmax, 12-14 of RPE) aerobic treadmill walking, 40 minutes including warm-up and cool-down times] , and the high-intensity interval exercise (HIIT) program with EX1 [High-intensity-low-intensity interval walking exercise was performed at treadmill speed (High: 90-95% HRmax, 15-17 of RPE/Low: 60-70% HRmax, 9-11 of RPE) and EX1 resistance strength (High: resistance intensity 7- 9/Low: Resistance strength 0-2)] to check the effect on muscle activity, heart rate, and respiratory metabolic energy consumption rate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 65 years without a history of central nervous system disease

Exclusion Criteria:

* Those who have difficulty walking independently due to problems such as visual field defects or fractures
* Those who have difficulty understanding the exercise program due to severe cognitive decline (Korean-Mini-Mental State Examination, K-MMSE≤10)
* Those who have difficulty participating in exercise programs due to adult diseases such as uncontrolled hypertension and diabetes
* Those who are at risk of falling while walking due to severe dizziness
* Those who are less than 140 cm or more than 185 cm in height that is not suitable size for the wearing of the walking assistance robot
* Those who are overweight based on body mass index (BMI) 35 or higher

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal adults aged 19 to 65 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Reduction on muscle activity (%MVC) | 3hours/2hours
  [aerobic] All subjects underwent measurements of the trunk and lower extremity muscle activity (%MVC) during aerobic treadmill walking and measured by three conditions (①Aerobic treadmill walking program without EX1, ②Aerobic treadmill walking program with EX1, and ③High-intensity interval exercise (HIIT) program with EX1.
  [anaerobic] All subjects underwent measurements of the trunk and lower extremity muscle activity (%MVC) during each condition

SECONDARY OUTCOMES:
Reduction on metabolic energy expenditure (ml·kg-1·min-1) | 3hours
  [aerobic] All subjects underwent measurements of respiratory metabolism energy (ml·kg-1·min-1) during aerobic treadmill walking and measured by three conditions (①Aerobic treadmill walking program without EX1, ②Aerobic treadmill walking program with EX1, and ③High-intensity interval exercise (HIIT) program with EX1.
Reduction on heart rate (beats per minute, bpm) | 3hours
  [aerobic] All subjects underwent measurements of heart rate (bpm) during aerobic treadmill walking and measured by three conditions (①Aerobic treadmill walking program without EX1, ②Aerobic treadmill walking program with EX1, and ③High-intensity interval exercise (HIIT) program with EX1.
Distinction on muscle activity (%MVC) | 3hours
  [aerobic] Exercising with EX1 results in higher muscle activity than exercising without wearing EX1.
Distinction on metabolic energy expenditure (ml·kg-1·min-1) | 3hours
  [aerobic] Exercising with EX1 consumes more energy for the same amount of time than exercising without wearing EX1.
Distinction on heart rate (beats per minute, bpm) | 3hours
  [aerobic] Exercising with EX1 shows a higher heart rate for the same time than exercising without EX1.
Distinction on muscle activity (%MVC) | 2hours
  [anaerobic] Fitness movements using EX1 generate more muscle activity than exercise without EX1.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea